CLINICAL TRIAL: NCT02729467
Title: An Open-Label Fixed-Sequence Study to Assess the Effects of Itraconazole and Rifampicin on the Single-Dose Pharmacokinetics of JNJ-53718678 in Healthy Adult Subjects
Brief Title: A Study to Assess the Effects of Itraconazole and Rifampicin on the Single-Dose Pharmacokinetics of JNJ-53718678 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108127; 53718678RSV1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2016-03-18; First posted 2016-04-06 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; JNJ-53718678; Itraconazole; Rifampicin; Pharmacokinetics
MeSH Terms: interventions — JNJ-53718678; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Panel 1 (Experimental): Participants will receive a single 250 milligram (mg) dose of JNJ-53718678 on Day 1 and 200 mg itraconazole once a day on Days 4 to 11 along with a single 250-mg dose of JNJ-53718678 on Day 9.
  Interventions: Drug: JNJ-53718678; Drug: Itraconazole
- Panel 2 (Experimental): Participants will receive a single 500-mg dose of JNJ-53718678 on Day 1; a single 600-mg dose of rifampicin along with a single 500-mg dose of JNJ-53718678 on Day 4 and 600 mg rifampicin once daily on Days 5 to 11 along with a single 500-mg dose of JNJ-53718678 on Day 9.
  Interventions: Drug: JNJ-53718678; Drug: Rifampicin

INTERVENTIONS:
Drug: JNJ-53718678 — JNJ-53718678 will be applied twice at doses of 250 mg (in Panel 1, Day 1 and Day 9) and 3 times at 500 mg (Panel 2, Day 1, 4 and 9).
Drug: Itraconazole — Participants will receive itraconazole 200 mg (2 capsules of 100 mg) from Day 4-11.
  Arms: Panel 1
Drug: Rifampicin — Participants will receive 600 mg rifampicin (2 capsules of 300 mg) from Day 4-11.
  Arms: Panel 2

SUMMARY:
The purpose of this study is to assess the effects of itraconazole, a strong cytochrome P (CYP)3A4 and p-glycoprotein (PgP) inhibitor, and rifampicin, a CYP3A4, uridine 5'-diphospho-glucuronosyltransferase (UGT), and PgP inducer, and an inhibitor of organic anion-transporting polypeptide (OATP), on the single-dose pharmacokinetics (PK) of JNJ-53718678 in healthy adult participants.

DETAILED DESCRIPTION:
This is a single-center, open-label, fixed sequence, Phase 1 study in healthy adult participants to study the effects of itraconazole and rifampicin on the pharmacokinetics, safety, and tolerability of a single dose of JNJ-53718678. This study will be conducted in 2 separate panels, with 14 participants in Panel 1 and 16 participants in Panel 2. The study consists of following phases: Screening (28 days), Treatment phase (11 days) and Follow-up (10 to 14 days after the last study drug intake). Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Participants will be assessed for safety and tolerability throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participants must have a negative serum beta human chorionic gonadotropin (beta hCG) pregnancy test at Screening
* At Screening, a female participant must be of non-childbearing potential
* Participant must have a Body Mass Index (BMI; weight in kilogram (kg) divided by the square of height in meters) of 18.0 to 30.0 kilogram per meter square (kg/m2), extremes included
* Participant must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and not higher than 90 mm Hg diastolic
* Participants must be healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination (including height and body weight measurement and skin examination), medical history, vital signs, and the results of blood biochemistry, blood coagulation, and hematology tests, and a urinalysis performed at Screening

Exclusion Criteria:

* Participant with a history of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic insufficiency, renal dysfunction, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participants with abnormal values for alanine aminotransferase (ALT) and aspartate aminotransferase (AST) (greater than [>]1.00 * upper limit of laboratory normal range [ULN])
* Participants with lack of good/reasonable venous access
* Participants with a past history of heart arrhythmias (extrasystoli, tachycardia at rest) or, history of risk factors for Torsade de Pointes syndrome (example - hypokalemia, family history of long QT Syndrome)
* Participants with any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) | Up to 11 days
  The Cmax is the maximum observed analyte concentration after the JNJ-53718678 doses on Day 1, Day 4 (Panel 2 only) and Day 9.
Area Under the Analyte Concentration-Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUC [0-last]) | Up to 11 days
  The (AUC [0-last]) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration after the JNJ-53718678 doses on Day 1 and Day 9.
Area Under the Analyte Concentration-Time Curve From Time 0 to Infinite Time (AUC [0-infinity]) | Up to 11 days
  The AUC (0-infinity) is the area under the Analyte concentration-time curve from time 0 to infinite time after the JNJ-53718678 doses on Day 1 and Day 9, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentrations; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Analyte Concentration-time curve From Time 0 to 24h (AUC24h) | Up to 11 days
  The AUC24h is the area under the analyte concentration-time curve from time 0 to 24h after dosing on Day 1 and Day 4 (Panel 2 only).
Ratio of Individual Cmax Values Between Test and Reference Treatment (Ratio Cmax, test/reference) | Up to 11 days
  Ratio Cmax, test/reference is the ratio of individual Cmax values between test (JNJ-53718678 with itraconazole, on Day 9, or JNJ-53718678 with rifampicin, on Day 4 and Day 9) and reference (without itraconazole or rifampicin, on Day 1) treatments.
Ratio of Individual AUC24h Values Between Test and Reference Treatment (Ratio AUC24h, test/reference) | Up to 11 days
  Ratio AUC24h, test/reference is the ratio of individual AUC24h values between test (JNJ-53718678 with rifampicin, on Day 4) and reference (without rifampicin, on Day 1) treatments.
Ratio of Individual AUClast Values Between Test and Reference Treatment (Ratio AUClast, test/reference) | Up to 11 days
  Ratio AUClast, test/reference is the ratio of individual AUClast values between test (JNJ-53718678 with itraconazole or rifampicin, on Day 9) and reference (without itraconazole or rifampicin, on Day 1) treatments.
Ratio of Individual AUC(infinity) Values Between Test and Reference Treatment (Ratio AUC[infinity], test/reference) | Up to 11 days
  Ratio AUC(infinity), test/reference is the ratio of individual AUC(infinity) values between test (JNJ-53718678 with itraconazole or rifampicin, on Day 9) and reference (without itraconazole or rifampicin, on Day 1) treatments.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events and Serious Adverse Events | Screening up to Follow-up (30 to 35 days after last study drug intake)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Overland Park, Kansas, United States